CLINICAL TRIAL: NCT00597103
Title: Comparison of Dialysis Therapies on Cognitive Function
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SR016CF
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease
Keywords: Hemodialysis; Frequent Hemodialysis; Sleep Apnea; Restless Leg Syndrome; Cognitive Function
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Sleep Apnea Syndromes; Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Prevalent patients who have been receiving more frequent dialysis.
  Interventions: Other: Cognitive Function Testing-10 Tests; Other: Sleep Assessment Testing; Other: Periodic Leg Movement Syndrome Assessment
- 2: Incident patients new to more frequent dialysis
  Interventions: Other: Cognitive Function Testing-10 Tests; Other: Sleep Assessment Testing; Other: Periodic Leg Movement Syndrome Assessment
- 3: Patients who switch from one more frequent hemodialysis treatment regimen to another more frequent dialysis regimen.
  Interventions: Other: Cognitive Function Testing-10 Tests; Other: Sleep Assessment Testing; Other: Periodic Leg Movement Syndrome Assessment

INTERVENTIONS:
Other: Cognitive Function Testing-10 Tests — Trailmaking A, Trailmaking B, Rey Auditory Verbal Learning, Letter Number Sequencing, Digit Symbol Substitution, Grooved Pegboard, Controlled Oral Word Association, Beck Depression Index, Feeling Thermometer, Modified Mini-Mental Status
Other: Sleep Assessment Testing — Sleep Assessment will be performed using an "Actiwatch" with subjects wearing the watch for 72 hours continuously
Other: Periodic Leg Movement Syndrome Assessment — Subjects will wear and "Actiwatch" on both legs for three consecutive nights.

SUMMARY:
This study will evaluate the effects of more frequent dialysis on cognitive function including the assessment of sleep apnea and restless legs. Our hypothesis is that more frequent dialysis improves cognitive function and may have important implications on clinical care of ESRD patients and help to emphasize the need for treatments that will allow patients to live "with dialysis" rather than live "for dialysis".

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ESRD
* Age 18 years or greater
* Ability to understand and a willingness to sign an informed consent statement and a Health Insurance Portability and Accountability Act of 1996 (HIPPA) authorization statement.
* Expected survival of at least one year.

Exclusion Criteria:

* Documented non-compliance, defined as missing more than 10% of prescribed treatments during the month prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Chronic Kidney Disease (CKD) who require renal replacement therapy and who are currently receiving dialysis.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04-05 (Actual); Study Completion 2011-04-05 (Actual)

PRIMARY OUTCOMES:
Distribution of cognitive function impairment in ESRD patients undergoing more frequent hemodialysis | baseline, 4 months and 12 months

SECONDARY OUTCOMES:
Longitudinal analysis of cognitive function over time to test the hypothesis that more frequent hemodialysis contributes to delay in cognitive function impairment | baseline, 4 months and 12 months
To test the hypothesis that nightly or daily hemodialysis treatment can ultimately be proven to be cost effective options by preserving cognitive function. | 12 months
Influence of cognitive function on survival. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schiller-Moran, MD, Principal Investigator — Satellite Healthcare, Inc.
Locations (2):
- United States (2):
  - Satellite Healthcare, Inc, Mountain View, California
  - WellBound, Inc., Mountain View, California